CLINICAL TRIAL: NCT06770010
Title: Advancing Feasibility and Acceptability of Digital Cognitive Rehabilitation in Sickle Cell (ALL IN)
Brief Title: Advancing Feasibility and Acceptability of Digital Cognitive Rehabilitation in Sickle Cell Disease
Acronym: ALL IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Steven J. Hardy, Principal Investigator, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000906
Record Dates: First submitted 2024-01-04; First posted 2025-01-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cogmed+ (Experimental): Home-based digital cognitive rehabilitation and memory strategy training targeting working memory functioning.
  Interventions: Behavioral: Cogmed+

INTERVENTIONS:
Behavioral: Cogmed+ — Cogmed is a home-based, digital working memory training program compatible with tablet devices. The program, designed for children ages 7 and older, consists of engaging cognitive exercises that target skills involving visuospatial and verbal working memory. An essential component of Cogmed training involves assignment of an intervention "coach" who has access to detailed data on the user's training data. Families will have videoconference meetings once per week with an intervention coach to review progress, provide feedback and answer any questions that arise during treatment. In addition, participants' coaching calls will be supplemented with direct instruction on the use of memory strategies. Social support interventions will also be provided involving three primary approaches: (1) multi-family Cogmed Kickoff social events; (2) social incentives; and (3) peer navigator support.

SUMMARY:
This is a single site nonrandomized pilot clinical trial of the feasibility, acceptability, and efficacy of a combination treatment involving digital Cogmed working memory skills training, social support components, and memory strategy training to improve adherence to Cogmed in youth with sickle cell disease ages 7-16 years.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility of a novel approach to ameliorating cognitive deficits in children and adolescents with sickle cell disease (SCD). SCD is an understudied, life-limiting disease affecting 100,000 individuals in the United States and over 300,000 newborns globally every year. Youth with SCD are at substantial neurological risk given their increased likelihood of overt stroke and silent cerebral infarct. However, even individuals without signs of cerebral infarct exhibit lower cognitive performance compared to healthy siblings due in large part to non-stroke, disease effects on the central nervous system. Disease-related cognitive issues are diffuse but often affect working memory function. Very few studies have examined therapeutic approaches to treating cognitive deficits in SCD; however, recent research supports the use of a home-based, eHealth working memory training program (Cogmed). In a randomized controlled trial, Cogmed training (i.e., repeated and adaptive working memory skills practice) resulted in improved working memory but adherence to the intervention was low. Early engagement with the training program emerged as predictive of better adherence. Therefore, in an effort to promote engagement, an enhanced version of the program was developed that incorporates social support components (e.g., multifamily Cogmed Kickoff events, social incentives, peer navigator support) and memory strategy training. The study will evaluate the following specific aims in a single-arm pilot clinical trial: 1) Assess the feasibility of Cogmed+ (Cogmed plus social support components and memory strategy training) in youth with SCD; and 2) Determine the effect of Cogmed+ on rates of treatment adherence. In this study, 50 youth ages 7-16 with SCD will complete a cognitive screening, after which 30 participants with working memory deficits will proceed to the Cogmed+ program. Participants will complete Cogmed on a tablet device from home 3-5 times per week for 5-8 weeks. Participants will attend weekly videoconference calls with a Cogmed coach who will review training progress and teach memory strategies during four coaching calls (weeks 2-5). Outcomes will be assessed by examining the number of Cogmed sessions completed and rates of attendance to Cogmed Kickoff events and memory strategy training sessions. Results will also be compared to a historical comparison group of youth with SCD who completed the basic version of Cogmed. Findings will provide critical data regarding a novel strategy for improving access to an efficacious treatment for youth with SCD. If such an augmented approach proves beneficial, resultant data will inform a randomized controlled trial to examine the effectiveness of a stepped care model that selectively delivers more intensive Cogmed treatment packages only as needed. This line of investigation, which balances practical access and resource considerations, could serve as a scalable care model and ignite efforts to address SCD-related cognitive impairment for the millions of people living with SCD globally.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell disease (any genotype).
2. Between ages 7-16 years old.
3. Patients will only enter the treatment phase if they score >1 SD below the normative mean on at least one standardized working memory assessment (i.e., Digit Span or Spatial Span subtests) or demonstrate a relative weakness in working memory (>1 SD below the estimated IQ).

Exclusion Criteria:

1. Motor, visual, or auditory impairment that prevents computer use.
2. Diagnosis of a mental health condition that precludes, or takes treatment precedence over, participation in the cognitive training.
3. History of photosensitive seizures.
4. Insufficient English fluency.
5. Recent initiation or dose adjustment of a stimulant medication to treat attention problems (< 30 days).

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete Cogmed training | Approximately 5-8 weeks after start of Cogmed training
  At least 75% of participants will complete 10 or more Cogmed training sessions.
Number of participants who attend a Cogmed Kickoff social event | Within approximately 6 months of study enrollment
  At least 75% of participants will attend a Cogmed Kickoff social event.
Number of participants who participate in memory strategy training | Approximately 5-8 weeks after start of Cogmed training
  At least 75% of participants will complete 2 or more memory strategy training sessions.

SECONDARY OUTCOMES:
Number of Cogmed training sessions completed | Approximately 5-8 weeks after start of Cogmed training
  Participants receiving the enhanced Cogmed intervention (including memory strategy training and social support components) will complete significantly more cognitive training sessions than a historic cohort who received Cogmed only.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hardy, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No